CLINICAL TRIAL: NCT01311921
Title: The Specific Aims Are to Find Factors Associated With Different Severe/Fatal Incidences in Different Areas of Taiwan. We Will do 1. Comparison of Gene Variants in EV71 Cases With Different Severity and Normal Children in Different Areas of Taiwan to Find Susceptible Genes and Genetic Polymorphism Related to the Clinical Outcomes 2. Social, Behavioral and Environmental Factors Related to EV71 Infections in Different Areas of Taiwan
Brief Title: Children's Susceptibility to Enterovirus 71 in Different Areas of Taiwan
Acronym: DMR100-IRB-010
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: China Medical University Hospital (Other)
Responsible Party: Kao-Pin,Hwang/Director of Pediatric Infectious Diseases, China Medical University Hospital
Other Study IDs: ChinaMUH
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Enterovirus 71, Host Genetics, Social, Behavior, Environmental Factors
Keywords: enterovirus 71, host genetics, social, behavior, environmental factors
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA,swab,blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
EV71 has caused large epidemics with lots of fatal cases and cases with sequelae. However, the clinical syndromes and severity of the same EV71 strain are very diverse, ranging from asymptomatic (71%) to fatal (0.05%) disease, and the pathogenesis remains unknown. In addition, the severe or fatal case incidence varies significantly differently in different areas of Taiwan. Although some viral virulence studies were performed, no clear viral virulence factor has been found. Therefore, host factors may be important to the clinical outcomes of EV71 infections. In addition, there were significantly different incidences of severe or fatal cases in different areas of Taiwan, for example, significantly more fatal or severe cases occurred in the central or southern Taiwan in comparison with in northern Taiwan. Whether this is related to host factors, social, behavioral or environmental factors remains unanswered. To find the most important factors associated with EV71 susceptibility, a thorough study involving genetics, social, behavioral or environmental factors among different areas of Taiwan is warranted and the findings will provide future prevention of EV71 and give help on early precaution and treatment of EV71.

DETAILED DESCRIPTION:
The specific aims are to find factors associated with different severe/fatal incidences in different areas of Taiwan. We will do

1. Comparison of gene variants in EV71 cases with different severity and normal children in different areas of Taiwan to find susceptible genes and genetic polymorphism related to the clinical outcomes
2. Social, behavioral and environmental factors related to EV71 infections in different areas of Taiwan

ELIGIBILITY:
Inclusion Criteria:

- Enterovirus type 71

Exclusion Criteria:

- not Enterovirus type 71

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Symptoms very like Enterovirus type 71 of hand, foot, and mouth disease or Herpangina,
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02